CLINICAL TRIAL: NCT05621174
Title: The Difference in Pharmacodynamic and Pharmacokinetic Profiles Between Tentin and Magisterial Dexamfetamine in Adults With Attention Deficit Hyperactivity Disorder, a Double Blinded Randomised Crossover-controlled Trial
Brief Title: The Difference in the Mechanism of Action Between Two Brands of Dexamfetamine in Adults With ADHD
Acronym: DAVE
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Responsible Party: Principal Investigator, Glenn Dumont, Associate professor, Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Other
Other Study IDs: 82695; 2022-003237-19 (EudraCT Number); 82695 (Registry Identifier: Centrale Commissie Mensgebonden Onderzoek (CCMO))
Record Dates: First submitted 2022-11-04; First posted 2022-11-17 (Actual); Last update posted 2025-02-18 (Actual); Status verified 2025-02

CONDITIONS: Attention Deficit Disorder With Hyperactivity
Keywords: Attention Deficit Disorder with Hyperactivity; Attention Deficit Hyperactivity Disorder; ADHD; ADD; AD(H)D
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity | interventions — Dextroamphetamine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Magisterial Dexamphetamine (Other): Magisterial Dexamphetamine
  Interventions: Drug: Dexamfetamine
- Tentin (Other): Tentin
  Interventions: Drug: Dexamfetamine

INTERVENTIONS:
Drug: Dexamfetamine — Magisterial Dexamfetamine
  Other Names: Magisterial Dexamfetamine
  Arms: Magisterial Dexamphetamine
Drug: Dexamfetamine — Tentin
  Other Names: Tentin
  Arms: Tentin

SUMMARY:
The goal of this clinical trial is to compare in the pk/pd profiles of magisterial dexamfetamine and Tentin in adults with Attention Deficit Hyperactivity Disorder (ADHD). The main question[s] it aims to answer are:

Q1: is there a difference between pk/pd profiles of the two forms of dexamfetamine?

Q2: how does the pharmacokinetic variability influences the objective and subjective (side) effects experienced by adult patients with ADHD?

Participants will:

* take the Quantified behavior Test for analysis of objective effects.
* undergo blood sampling for analysis of the plasma concentration of dexamphetamine.
* undergo blood pressure and heart rate measurements.
* fill out 4 types of questionnaires.

Researchers will compare the outcomes between magisterial dexamphetamine and Tentin use in a crossover setting.

DETAILED DESCRIPTION:
Objectives The primary objective is to compare the pharmacological profile of the magisterial form of dexamfetamine sulfate to the pharmacological profile of the brand-name form of dexamfetamine (Tentin©) in adult patients diagnosed with attention deficit hyperactivity disorder (ADHD) and assess whether there is a difference between pk/pd profiles of the two forms of dexamfetamine. The secondary objective is to assess how pharmacokinetic variability influences the objective and subjective (side) effects experienced by adult patients with ADHD.

Measurements At three moments (0, 60 and 120 minutes after drug administration) on each intervention-day, participants will complete the QbTest to assess objective performance and the QbPerformance to assess subjective performance. At eight moments (0, 45, 60, 75, 90, 120, 150 and 180 minutes after drug administration) on each intervention-day, participants will undergo blood sampling to determine dexamfetamine plasma concentrations and vital sign measurements for safety monitoring and possible outcome-effects. At eight moments (0, 45, 60, 75, 90, 120, 150 and 180 minutes after drug administration) on each intervention-day, participants will fill out questionnaires to assess subjective experiences.

ELIGIBILITY:
Inclusion Criteria:

* Participant is aged ≥ 18 years at time of screening.
* Participant is diagnosed with ADHD according to the DSM 5 criteria.
* Participant has switched from Tentin© to magisterial dexamfetamine due to the adverse effects of Tentin.
* Participant is being treated adequately with dexamphetamine, as determined by their practitioner, at time of screening.
* Participant or their legal representative is able and willing to provide written informed consent.
* Participant is able and willing to comply with the study protocol (e.g. swallow capsules, have blood samples taken, can visit the outpatient clinic twice).
* Participant has not participated in another study in the past three months.

Exclusion Criteria:

* Participant has a disorder that might affect drug absorption (e.g. gastrointestinal, metabolic, endocrine or liver disorder).
* Participant is allergic to the ingredients of the capsules.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 1 (Actual)
Dates: Start 2023-04-14 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Quantified behavior Test (QbTest) - Time Active | 0-120 minutes after drug administration
  Time Active for analysis of objective effects. The Quantified behaviour Test (QbTest) provides data to assess the three core symptoms of ADHD, that is: hyperactivity, inattention and impulsivity. Time Active (in %) is one of the scores used to measure hyperactivity, inattention and impulsivity. For the current study cardinal outcomes will be derived from a Principal Component Analysis.
Quantified behavior Test (QbTest) - Distance | 0-120 minutes after drug administration
  Distance for analysis of objective effects. The Quantified behaviour Test (QbTest) provides data to assess the three core symptoms of ADHD, that is: hyperactivity, inattention and impulsivity. Distance (in meters) is one of the scores used to measure hyperactivity, inattention and impulsivity. For the current study cardinal outcomes will be derived from a Principal Component Analysis.
Quantified behavior Test (QbTest) - Area | 0-120 minutes after drug administration
  Area for analysis of objective effects. The Quantified behaviour Test (QbTest) provides data to assess the three core symptoms of ADHD, that is: hyperactivity, inattention and impulsivity. Area (in cm2) is one of the scores used to measure hyperactivity, inattention and impulsivity. For the current study cardinal outcomes will be derived from a Principal Component Analysis.
Quantified behavior Test (QbTest) - Micro Events | 0-120 minutes after drug administration
  Micro Events for analysis of objective effects. The Quantified behaviour Test (QbTest) provides data to assess the three core symptoms of ADHD, that is: hyperactivity, inattention and impulsivity. Micro Events (in millimeters) is one of the scores used to measure hyperactivity, inattention and impulsivity. For the current study cardinal outcomes will be derived from a Principal Component Analysis.
Quantified behavior Test (QbTest) - Motion Simplicity | 0-120 minutes after drug administration
  Motion Simplicity for analysis of objective effects. The Quantified behaviour Test (QbTest) provides data to assess the three core symptoms of ADHD, that is: hyperactivity, inattention and impulsivity. Motion Simplicity (in %) is one of the scores used to measure hyperactivity, inattention and impulsivity. For the current study cardinal outcomes will be derived from a Principal Component Analysis.
Blood samples | 0-180 minutes after drug administration
  For analysis of the plasma concentration of dexamfetamine.
Blood pressure | 0-180 minutes after drug administration
  For autonomic and adverse effects measurements. Measured in mmHg Normal value: 120/80 mmHg
Heart rate | 0-180 minutes after drug administration
  For autonomic and adverse effects measurements. Measured in BPM Normal value: 60-100 BPM

SECONDARY OUTCOMES:
Addiction Research Centre Inventory (ARCI) - Acute Subjective Response to Substances (ASRS): Amphetamine Scale | 45-180 minutes after drug administration
  Subjective effects measurement In this trial, only amphetamines will be administered, therefore only the first 11 questions of the amphetamine-scale will be used. The investigators have adjusted the 'true-false' questions in the amphetamine-scale to Visual Analog Scale (VAS)-questions, since VASs are more sensitive to subtle changes than Likert-scales and VAS enables rapid completion leading to a lower participant burden. The ARCI questions 1 t/m 11 are in line with the therapeutic effects of dexamfetamine.
  For each question, the VAS can be marked between 0 and 10 cm, 0 meaning 'not at all' and 10 meaning 'very much' when answering the questions.
Bond-Lader Visual Analog Scale (BL-VAS) | 0-180 minutes after drug administration
  Subjective effects measurement The Bond & Lader VAS Mood Rating Scale (BL-VAS) is used to measure the effects of drugs on the participants' mood. It consists of 16 dimensions (VAS) of mood. Ultimately, these dimensions are combined to create the following dimensions: alertness, contentedness, and calmness.
  For each question, the VAS can be marked between 0 and 10 cm, 0 meaning 'not at all' and 10 meaning 'very much' when answering the questions.
QbTest performance questionnaire | 0-180 minutes after drug administration
  Subjective effects measurement QbPerformance to assess subjective performance on the QbTest.
  For 1 question, a 'yes' or 'no' answer will be given. For 3 questions, the VAS can be marked between 0 and 10 cm, 0 meaning 'not at all' and 10 meaning 'very much' when answering the questions.

OTHER OUTCOMES:
Leeds Sleep Evaluation Questionnaire (LSEQ) | Before drug administration
  Sleep deprivation can negatively impact attention functioning in adults with and without ADHD. Sleep deprived participants performed worse on the QbTest. Therefore, the sleep quality of participants must be taken into account. The Leeds Sleep Evaluation Questionnaire (LSEQ) consists of ten bipolar 100mm visual analogue scales (VAS) questions that are associated with sleep. The LSEQ covers the following four aspects of sleep, namely: getting to sleep, quality of sleep, awakening from sleep and behavior following wakefulness (F1-CRF). The LSEQ has provided evidence for validity in clinical research. Furthermore, the LSEQ has been cross-culturally validated in multiple countries and languages. The LSEQ is a consistent, reliable and validated tool to evaluate sleep and should therefore be included in the current study. Participants will be asked to fill in the questionnaire once at baseline (T=0), since it only evaluates the sleep quality of participants of the night before.

CONTACTS AND LOCATIONS:
Overall Officials: Glenn JH Dumont, PhD, Principal Investigator — Amsterdam UMC
Locations (1):
- Glenn Dumont, Amsterdam, North Holland, Netherlands

IPD SHARING:
Plan to Share IPD: No
Privacy protocol

REFERENCES:
- [Background] Lott DC, Kim SJ, Cook EH, de Wit H. Serotonin transporter genotype and acute subjective response to amphetamine. Am J Addict. 2006 Sep-Oct;15(5):327-35. doi: 10.1080/10550490600859868. PMID 16966188
- [Background] Martin WR, Sloan JW, Sapira JD, Jasinski DR. Physiologic, subjective, and behavioral effects of amphetamine, methamphetamine, ephedrine, phenmetrazine, and methylphenidate in man. Clin Pharmacol Ther. 1971 Mar-Apr;12(2):245-58. doi: 10.1002/cpt1971122part1245. No abstract available. PMID 5554941
- [Background] Wong YN, Wang L, Hartman L, Simcoe D, Chen Y, Laughton W, Eldon R, Markland C, Grebow P. Comparison of the single-dose pharmacokinetics and tolerability of modafinil and dextroamphetamine administered alone or in combination in healthy male volunteers. J Clin Pharmacol. 1998 Oct;38(10):971-8. doi: 10.1002/j.1552-4604.1998.tb04395.x. PMID 9807980
- [Background] Dolder PC, Strajhar P, Vizeli P, Hammann F, Odermatt A, Liechti ME. Pharmacokinetics and Pharmacodynamics of Lisdexamfetamine Compared with D-Amphetamine in Healthy Subjects. Front Pharmacol. 2017 Sep 7;8:617. doi: 10.3389/fphar.2017.00617. eCollection 2017. PMID 28936175
- [Background] Dan O, Cohen A, Asraf K, Saveliev I, Haimov I. The Impact of Sleep Deprivation on Continuous Performance Task Among Young Men With ADHD. J Atten Disord. 2021 Jul;25(9):1284-1294. doi: 10.1177/1087054719897811. Epub 2020 Jan 9. PMID 31916494
- [Background] Parrott AC, Hindmarch I. The Leeds Sleep Evaluation Questionnaire in psychopharmacological investigations - a review. Psychopharmacology (Berl). 1980;71(2):173-9. doi: 10.1007/BF00434408. PMID 6777817
- [Background] Tarrasch R, Laudon M, Zisapel N. Cross-cultural validation of the Leeds sleep evaluation questionnaire (LSEQ) in insomnia patients. Hum Psychopharmacol. 2003 Dec;18(8):603-10. doi: 10.1002/hup.534. PMID 14696019
- [Background] Manzar MD, Salahuddin M, Maru TT, Alghadir A, Anwer S, Bahammam AS, Pandi-Perumal SR. Validation of the adapted Leeds sleep evaluation questionnaire in Ethiopian university students. Health Qual Life Outcomes. 2018 Mar 13;16(1):49. doi: 10.1186/s12955-018-0876-0. PMID 29534726
- [Background] Haertzen CA. Development of scales based on patterns of drug effects, using the addiction Research Center Inventory (ARCI). Psychol Rep. 1966 Feb;18(1):163-94. doi: 10.2466/pr0.1966.18.1.163. No abstract available. PMID 5908477
- [Background] HILL HE, HAERTZEN CA, WOLBACH AB Jr, MINER EJ. THE ADDICTION RESEARCH CENTER INVENTORY: STANDARDIZATION OF SCALES WHICH EVALUATE SUBJECTIVE EFFECTS OF MORPHINE, AMPHETAMINE, PENTOBARBITAL, ALCOHOL, LSD-25, PYRAHEXYL AND CHLORPROMAZINE. Psychopharmacologia. 1963 May 15;4:167-83. doi: 10.1007/BF02584089. No abstract available. PMID 14048539
- [Background] Lader MH, Bond AJ. Interaction of pharmacological and psychological treatments of anxiety. Br J Psychiatry Suppl. 1998;(34):42-8. PMID 9829016
- [Background] Setnik B, Roland CL, Pixton G, Webster L. Measurement of Drug Liking in Abuse Potential Studies: A Comparison of Unipolar and Bipolar Visual Analog Scales. J Clin Pharmacol. 2017 Feb;57(2):266-274. doi: 10.1002/jcph.801. Epub 2016 Aug 23. PMID 27444046
- [Background] Ahearn EP. The use of visual analog scales in mood disorders: a critical review. J Psychiatr Res. 1997 Sep-Oct;31(5):569-79. doi: 10.1016/s0022-3956(97)00029-0. PMID 9368198
- [Background] Ashinoff BK, Abu-Akel A. Hyperfocus: the forgotten frontier of attention. Psychol Res. 2021 Feb;85(1):1-19. doi: 10.1007/s00426-019-01245-8. Epub 2019 Sep 20. PMID 31541305
- [Background] Schmid Y, Hysek CM, Simmler LD, Crockett MJ, Quednow BB, Liechti ME. Differential effects of MDMA and methylphenidate on social cognition. J Psychopharmacol. 2014 Sep;28(9):847-56. doi: 10.1177/0269881114542454. Epub 2014 Jul 22. PMID 25052243
- [Background] Pourhoseingholi MA, Baghestani AR, Vahedi M. How to control confounding effects by statistical analysis. Gastroenterol Hepatol Bed Bench. 2012 Spring;5(2):79-83. PMID 24834204
- [Background] Kang H. The prevention and handling of the missing data. Korean J Anesthesiol. 2013 May;64(5):402-6. doi: 10.4097/kjae.2013.64.5.402. Epub 2013 May 24. PMID 23741561
- See also: Summary of Product Characteristics - DMB 5 mg — https://www.geneesmiddeleninformatiebank.nl/smpc/h115446_smpc.pdf
- See also: Summary of Product Characteristics - Tentin 5 mg — https://www.geneesmiddeleninformatiebank.nl/smpc/h124800_smpc.pdf